**Statistical Analysis Plan Template** 

**BI Study Number 1237-0070.** 

Protocol Version 1.0. Date: 19 September 2017

Non-interventional, cross-sectional, multicenter study to describe the exacerbations profile of COPD patients Treated with ICS in a real-life primary care population in Spain. OPTI Study.

**Author:** 

Version Number and Date: V1.0; 29 May 2019

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx

Author: Version Number: 1.0

Version Date: [29MAY2019]

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 

#### STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

# Statistical Analysis Plan <V1.0, 29 MAY 2019)> for Protocol 1237-0070.

| | Name | Signature | Date |
|--------------|-----------------|-----------|------|
| Author: | | | |
| Position: | Statistician | | |
| Company: | | | |
| | Name | Signature | Date |
| Approved By: | | | |
| Position: | Project | <u> </u> | ' |
| Company: | | | |
| Approved By: | | | |
| Position: | Medical Project | | |
| Company: | | | |
| Approved By: | | | |
| Position: | Statistician | | |
| Company: | | | |
| | · | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

## MODIFICATION HISTORY

| Unique Identifier | Date of the | Author | Significant Changes from |
|-------------------|-------------|--------|------------------------------|
| for this Version | Document | | Previous Authorized Version |
| | Version | | |
| 0.1 | 20-JUL-2018 | | Not Applicable – First draft |
| 0.2 | 20-FEB-2019 | | No |
| 0.3 | 18-MAR-2019 | | No |
| 0.4 | 24-APR-2019 | | No |
| 0.5 | 07-MAY-2019 | | No |
| 0.6 | 08-MAY-2019 | | No |
| 0.7 | 21-MAY-2019 | | No |

 $\label{thm:constraint} $$ \c SO_{\c SO_2017 \ actualizada}. SRO\ ESTUDIOS\RESPIRATORIO\1237-0070\ NISO_{\c SO_2017 \ actualizad$ Document:

Version Number: Author: 1.0


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

## TABLE OF CONTENTS

| 1. | ABB | REVIAT | ONS | 8 |
|---|---|---|---|---|
| 2. | INT | RODUCT | ION | 9 |
| 3. | STU | DY OBJE | CTIVES | 9 |
| | 3.1 | Primary | Objective | 9 |
| | 3.2 | Seconda | ary Objectives | 9 |
| 4. | STU | DY DESI | GN | 10 |
| | 4.1 | General | Description | 10 |
| | 4.2 | Study si | ze | 10 |
| | 4.3 | Descrip | tion of the treatment | 11 |
| | 4.4 | Study fl | ow/schedule | 11 |
| | 4.5 | Schedul | e of Events | 12 |
| | 4.6 | Change | s to Analysis from Protocol | 12 |
| <b>5.</b> | PLA | NNED AN | NALYSES | 12 |
| | 5.1 | Interim | Analysis | 12 |
| | 5.2 | Final A | nalysis | 12 |
| 6. | ANA | LYSIS SI | ETS | 13 |
| | 6.1 | Subjects | s enrolled (ENR) | 13 |
| | 6.2 | Full An | alysis Set (FAS) | 13 |
| | 6.3 | Patients | treated with ICS Analysis Set (PICAS) | 14 |
| | 6.4 | Safety A | Analysis Set - ICS | 14 |
| | 6.5 | | Analysis Set - SPIOLTO®, STRIVERDI®, SPIRIVA® or /ENT® | 14 |
| 7. | GEN | ERAL CO | ONSIDERATIONS | 14 |
| | 7.1 | Referen | ce Start/End Date | 15 |
| | 7.2 | Commo | n Calculations | 15 |
| | | 7.2.1 | Body Mass Index (BMI) | 15 |
| | | 7.2.2 | Number of Pack-years | 16 |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Template No.: RWI\_TP\_BIOS0013 Revision 1

| | | 7.2.3 | Time since COPD diagnosis | 16 |
|---|---|---|---|---|
| | | 7.2.4 | Time since Asthma diagnosis | 16 |
| | | 7.2.5 | Spirometric values | 16 |
| | | 7.2.6 | Number of exacerbations | 17 |
| | | 7.2.7 | Laboratory values | 17 |
| | | 7.2.8 | GOLD 2019 | 18 |
| | | 7.2.9 | BODEx Index | 18 |
| | | 7.2.10 | COTE Index | 19 |
| | | 7.2.11 | Risk stratification | 20 |
| | | 7.2.12 | Gold 2019 Classification | 21 |
| | | 7.2.13 | CAT questionnaire score | 21 |
| | | 7.2.14 | Adherence to ICS treatment recommendations according GesEPOC 2017 guideline. | 22 |
| | 7.3 | Software | Version | 25 |
| 8. | STAT | ISTICAL | CONSIDERATIONS | 25 |
| | 8.1 | Statistica | l Bias Reduction | 25 |
| | 8.2 | Statistica | l Tests and Confidence Intervals | 25 |
| | 8.3 | Adjustme | ents for Covariates and Factors to be Included in Analyses | 26 |
| | 8.4 | Missing of | data | 26 |
| 9. | OUTI | PUT PRES | SENTATIONS | 27 |
| 10. | DISPO | OSITION | AND WITHDRAWALS | 28 |
| 11. | DEM | OGRAPH | IC AND OTHER BASELINE CHARACTERISTICS | 28 |
| | 11.1 | Derivatio | ons | 28 |
| 12. | SURC | GICAL AN | ND MEDICAL HISTORY | 28 |
| 13. | COM | ORBIDIT | TES | 28 |
| 14. | MED | ICATION | S | 29 |
| 15. | STUD | Y MEDIO | CATION EXPOSURE | 29 |
| 16. | PRIMARY OUTCOMES | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

| | 16.1 | Primary | Endpoint | 29 |
|---|---|---|---|---|
| | | 16.1.1 | Data Variables and Derivation | 29 |
| | | 16.1.2 | Missing Data Methods for Primary Endpoint | 29 |
| | | 16.1.3 | Primary Analysis of Primary Endpoints | 30 |
| | 16.2 | Seconda | ry analysis | 32 |
| | | 16.2.1 | ICS use in the two years prior to the study visit | 32 |
| | | 16.2.2 | Moderate-to-severe exacerbations in COPD | 32 |
| | | 16.2.3 | General patient profile for COPD patients | 33 |
| | | 16.2.4 | Rescue medication use | 35 |
| | | 16.2.5 | Adherence to GesEPOC 2017 treatment recommendations guidelines | 35 |
| | | 16.2.6 | ICS-related adverse events | 36 |
| 17. | PATI | ENT REF | PORTED OUTCOMES (PRO) | 36 |
| 18. | SAFE | TY OUT | COMES | 36 |
| | 18.1 | Adverse | Drug Reactions | 36 |
| | 18.2 | Serious A | Adverse Drug Reactions | 37 |
| | 18.3 | Deaths | | 37 |
| 19. | REFE | ERENCES | S | 37 |
| | 19.1 | Dated & | Times | 38 |
| | 19.2 | Spelling | Format | 38 |
| | 19.3 | Listings. | | 38 |
| 20. | TABI | LES AND | FIGURES | 39 |
| | 20.1 | Evaluabi | ility | 39 |
| | 20.2 | General | patient profile for COPD patients according to ICS current use | 40 |
| | | 20.2.1 | Socio-demographic characteristics | 40 |
| | | 20.2.2 | Clinical variables | 42 |
| | | 20.2.3 | Exacerbations | 46 |
| | | 20.2.4 | Current COPD treatment. | 47 |
| | | 20.2.5 | Previous COPD treatment | 58 |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

| | 20.2.6 | Rescue medication | . 61 |
|---|---|---|---|
| | 20.2.7 | Concomitant treatments (ATC code classification) | . 63 |
| 20.3 | Endpoints | S | . 64 |
| | 20.3.1 | ICS treatment | . 64 |
| | 20.3.2 | Exacerbations | . 68 |
| | 20.3.3 | Adherence to treatment recommendations according GesEPOC 2017 guidelines. | 71 |
| 20.4 | Safety | | 72 |
| | 20.4.1 | Adverse Drug Reactions - related with ICS | . 72 |
| | 20.4.2 | Serious Adverse Drug Reactions (SADRs) - related with ICS | . 73 |
| | 20.4.3 | Adverse Drug Reactions associated to BI product (SPIOLTO®, STRIVERDI®, SPIRIVA® or ATROVENT®) | 74 |
| | 20.4.4 | Serious Adverse Drug Reaction (SADRs)related with BI product. | . 76 |
| | 20.4.5 | Deaths | . 77 |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

## 1. ABBREVIATIONS

ACOS Asthma COPD overlap syndrome

ADR Adverse Drug Reaction

AE Adverse Event

CI Confidence Interval

COTE Copd cO-morbidity Test

ENR Subjects enrolled

FEV<sub>1</sub> Forced expiratory volume in 1<sub>st</sub> second

FVC Forced vital capacity
ICS Inhaled corticosteroid
IgE Immunoglobulin E

ige illillulloglobulli e

LABA Long-acting beta2-agonist

mMRC Modified Medical Research Council

TLF Tables/Listings/Figures shells

SADR Serious Adverse Drug Reaction

SABA Short-acting beta2- agonists

SAMA Short-acting muscarinic antagonist

SAP Statistical Analysis Plan

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 

2. INTRODUCTION

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation

and analysis of treatment patterns and patient profile. It describes the data to be summarized and

analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 1.0, dated 19 September 2017 and

case report forms (CRFs) version 1.0, dated 28 June 2018.

3. STUDY OBJECTIVES

This study has been designed in order to describe the COPD patient profile of patients treated with or

without ICS in primary care, in Spain.

3.1 Primary Objective

The primary objective is to describe the patient profile for patients treated with ICS at the time of

study visit.

3.2 Secondary Objectives

The secondary objectives are:

To describe the patient profile for patients not treated with ICS at the time of study visit.

• To assess the proportion and the number (count) of patients with COPD treated with ICS at

the time of study visit with or without moderate-to-severe exacerbations, both in the previous

1 year and previous 2 years before the study visit.

• To assess the proportion and the number (count) of patients with COPD not treated with ICS

at the time of study visit with or without moderate-to-severe exacerbations, both in the

previous 1 year and previous 2 years before the study visit.

• Use of rescue medication.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

• Adherence to treatment recommendations according GesEPOC guidelines.

• To describe ICS-related adverse events.

4. STUDY DESIGN

4.1 General Description

This non-interventional, descriptive, cross-sectional cohort and multicentre study will be conducted

with COPD patients attended at Spanish Primary Care offices.

The design of the study imposes an only visit to be performed that will coincide with one of those

performed by the patients as part of routine follow-up of their disease, without interfering with usual

clinical practice of the investigator.

A specific therapeutic strategy has already been assigned to each included patient, based on routine

practice and without interference with the physician's prescription habits. The observational nature

of the study is ensured as no diagnostic or therapeutic intervention outside of routine clinical practice

will be applied.

4.2 Study size

Due to the descriptive design of the proposed non-interventional study, a formal sample size

calculation has not been performed based on statistical power and protection for type I error.

In previously published studies in Spain (Miravitlles, 2015), 66% of patients in usual clinical practice

attending to primary care are non-exacerbators and of these, 61% are treated with ICS, therefore

approximately 40% of all patients are currently treated with ICS without having exacerbations in the

prior year.

Assuming a sample size of 900 patients and 40% of the patients are treated with ICS at the study

visit and did not have a moderate or severe COPD exacerbation in the prior year, the 95% confidence

interval for this proportion would be between 36.8% (lower limit) and 43.2% (upper limit). To

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

account for a 10% drop-out rate (patients with inconsistent, incomplete or missing data), the sample size becomes 1,000 patients.

Table 1. Scenario for estimated proportions by 95% confidence intervals (95% CI)

| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
|---|---|---|---|---|---|---|---|---|
| Expected proportion | 0.4 | | | | 0.5 | | | |
| Lower and Upper limit of 95% CI | (0.37;0.43) | (0.368;0.432) | (0.365;0.435) | (0.363;0.437) | (0.47;0.53) | (0.468;0.532) | (0.465;0.535) | (0.463;0.537) |
| Precision of estimation | 0.030 | 0.032 | 0.035 | 0.037 | 0.030 | 0.032 | 0.035 | 0.037 |
| N (at final analysis) | 1000 | 900 | 753 | 674 | 1042 | 938 | 784 | 702 |
| Dropout 10% | 1112 | 1000 | 838 | 749 | 1159 | 1043 | 872 | 780 |

## 4.3 Description of the treatment

Patients in this study will have been prescribed a treatment for their COPD. They could have been prescribed ICS or not. Prescription of the treatments will have been done under the sole responsibility of the healthcare professional and before the study initiation visit.

In addition, no intervention, either diagnostic or therapeutic, will be applied to patients other than that used for routine clinical practice.

## 4.4 Study flow/schedule

The design of the study imposes only one visit to be performed that will coincide with one of those performed by the patients as part of routine follow-up of their disease, without interfering with usual clinical practice of the investigator.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 



Figure 1. Study scheme for study periods

After signing the informed consent (if patient agreed to participate in the study) patients will be asked to answer the breathlessness scale (mMRC) and the CAT – COPD Assessment Test at the unique study visit. Other variables needed to answer study objectives will be obtained directly from patient medical records. The end of the study visit is the end of the study for each patient.

#### 4.5 Schedule of Events

The schedule of events can be found in Section 6 of the protocol (Milestones).

## 4.6 Changes to Analysis from Protocol

No changes in analysis or definitions included in the final protocol have been considered.

## 5. PLANNED ANALYSES

## 5.1 Interim Analysis

No interim analysis has been planned.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

## 5.2 Final Analysis

All final, planned analyses identified in this SAP will be performed by

Real-World Evidence
Solutions (RWES) Biostatistics following

SOPs. Final CSR will be performed using
Boehringer Ingelheim template.

## 6. ANALYSIS SETS

## 6.1 Subjects enrolled (ENR)

Subjects enrolled (ENR) set will contain all subjects who provide informed consent for this study and are included in main database.

# 6.2 Full Analysis Set (FAS)

The Full Analysis Set (FAS) will contain all subjects who provide informed consent for this study (ENR set) and fulfill all selection criteria. To be eligible to participate in the study, patients must meet the following selection criteria. The patient will be considered included when he/she agrees to participate in the study by signing the informed consent. This analysis set includes patients fulfilling these conditions:

- 1) Written informed consent prior to participation.
- 2) Female and male patient  $\geq 40$  years of age.
- 3) COPD diagnosis more than 2 years before the study visit.
- 4) Previously confirmed COPD diagnosis (post-bronchodilator FEV1/FVC ratio <70%)
- 5) Clinical data available 2 years before the study visit.
- 6) Ability to complete CAT COPD Assessment Test.

Patients will be excluded from participating in this study, and will be excluded from this analysis set, if the following criterion is met:

1) Current participation in any clinical trial involving a drug or device.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

2) A moderate or severe exacerbation (requiring oral corticosteroid, antibiotics or hospitalisation) during the study visit or within 4 weeks before the study visit.

# 6.3 Patients treated with ICS Analysis Set (PICAS)

The patients treated with ICS Analysis Set (PICAS) includes all patient in FAS set treated with ICS during the study period.

## 6.4 Safety Analysis Set - ICS

The patients in the Safety Analysis Set includes all patient in ENR set treated at least with one dose of ICS during the study period. All safety variables related with ICS will be analyzed using this analysis set.

## 6.5 Safety Analysis Set - SPIOLTO®, STRIVERDI®, SPIRIVA® or ATROVENT®

The patients in the Safety Analysis Set includes all patient in ENR set treated at least with one dose of SPIOLTO®, STRIVERDI®, SPIRIVA® or ATROVENT® during the study period. All safety variables related to Boehringer Ingelheim COPD drugs will be analyzed using this analysis set.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

7. GENERAL CONSIDERATIONS

The design of the study imposes an only one visit to be performed that will coincide with one of

those performed by the patients as part of routine follow-up of their disease, without interfering with

usual clinical practice of the investigator.

Data will be obtained from patient medical records and during the study visit. Most of data will be

available in the charts but as a routine clinical practice, some data could be missing. Data will be

collected through an eCRF, which will include all the study variables.

The Investigator will enter the patient following the user guide during the study visit will fill in the

CAT – COPD Assessment Test and mMRC data electronically into the eCRF system.

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at

any time for the following reasons:

1. Failure to meet expected enrolment goals overall or at a particular study site

2. Emergence of any efficacy/safety information that could significantly affect continuation of the

study

3. Violation of the study protocol, or the contract by a study site or investigator, disturbing the

appropriate conduct of the study

7.1 Reference Start/End Date

Reference start date is date of study visit, collected in the eCRF as mandatory variable. For this

retrospective chart review study, index date is defined as date for data collection (patients attending

to the participant site).

Document:

\bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx

Author:

Version Number: 1.0


\_\_\_\_

Template No.: RWI\_TP\_BIOS0013 Revision 1

#### 7.2 Common Calculations

## 7.2.1 Body Mass Index (BMI)

The formula to obtain Body Mass Index is the following: BMI  $(kg/m^2)$  = weight (kg)/ height  $^2$  (m) and BMI will be categorized into 5 categories according to the World Health Organization (WHO):

• Underweight: BMI< 18.5 kg/m<sup>2</sup>

• Normal weight:  $18.5 \text{ kg m}^2 \le BMI \le 25 \text{ kg/m}^2$ 

• Overweight:  $25 \text{ kg/m}^2 < BMI <= 30 \text{ kg/m}^2$ 

• Obese:  $30 \text{ kg/m}^2 < \text{BMI} <= 35 \text{ kg/m}^2$ 

• Severely Obese: BMI> 35 kg/m<sup>2</sup>

# 7.2.2 Number of Pack-years

The number of **pack-years** is equal to the number of cigarettes smoked per day divided by 20 and multiplied by number of years smoked. The formula used for current smokers and ex-smokers will be:

Number of pack-years (for smokers) = (packs smoked per day) × (years smoking)

Number of pack-years (for Ex-Smokers) = (packs smoked per day)  $\times$  (years smoking)

# 7.2.3 Time since COPD diagnosis

The number of years since diagnosis will be obtained as the difference between year of study visit and year of COPD diagnosis (+1). Years since diagnosis could be categorized according quartiles (or percentiles).

#### 7.2.4 Time since Asthma diagnosis

In asthmatic patients, the number of years since diagnosis will be obtained as the difference between year of study visit and year of Asthma diagnosis (+1).

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

## 7.2.5 Spirometric values

Spirometric data are collected directly from clinical records. However, Predicted FEV<sub>1</sub>/FVC pre and post bronchodilator and change in FEV<sub>1</sub> will be calculated using the formulas:

```
Predicted FEV1 (L) = 100 x FEV1 (L) / FEV1 (%)

Predicted FVC (L) = 100 x FVC (L) / FVC (%)

Change (L) in FEV1 = FEV1 Post (L) - FEV1 Pre (L)

Percentage (1) of change in FEV1 (%) = 100 x [FEV1 Post (L) - FEV1 Pre (L)] / Predicted FEV1 (L)

Percentage (2) of change in FEV1 (%) = 100 x [FEV1 Post (L) - FEV1 Pre (L)] / Predicted FEV1 Pre (L)
```

#### 7.2.6 Number of exacerbations

## 7.2.6.1 Number of total exacerbations

The number of exacerbations (mild, moderate and severe) in the last two years will be the number of exacerbations registered in section 8 of CRF, whose date of exacerbation is included in the last 2 years or 730.50 days (365.25x2) before the study visit.

The number of exacerbations in the last year will be the number of exacerbations registered in section 8 of CRF, whose date of exacerbation is included in the last 365 days before the study visit.

In both cases, the number of exacerbations will be assumed as zero when "without exacerbation in the last 2 years" is ticked.

## 7.2.6.2 Number of severe exacerbations

The number of severe exacerbations in the last two years will be the number of exacerbations requiring hospitalization, registered in section 8 of CRF, whose date of exacerbation is included in the last 2 years or 730.5 days (365.25x2) before the study visit.

The number of severe exacerbations in the last year will be the number of exacerbations registered in section 8 of CRF, whose date of exacerbation is included in the last 365 days before the study visit and required hospitalization.

In both cases, the number of severe exacerbations will be assumed as zero when "without exacerbation in the last 2 years" is ticked.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

## 7.2.7 Laboratory values

## 7.2.7.1 Eosinophils

Eosinophils will be categorized in two categories (for each unit) (Celli 2017) (GOLD 2019):

- If eosinophils are in %: <2% and  $\ge 2\%$
- If eosinophils are in cells/ $\mu$ l: <100, 100-299 and  $\geq$ 300.

## 7.2.7.2 Immunoglobulin E

Immunoglobulin E (IgE) levels will be categorized according to these values, included in the Spanish Asthma guidelines (GEMA) and ACO (Cosio et al. 2016):

- <100 UI/ml
- >100 UI/ml

#### 7.2.8 GOLD 2019

To determine the severity of all subjects with COPD (independently of FEV<sub>1</sub>/FVC post-bronchodilation obtained), patients will be categorized into four levels, according to these criteria:

- Gold 1 (mild):  $FEV_1$  (%)>= 80% predicted.
- Gold 2 (Moderate): 50% <= FEV<sub>1</sub> (%) <80% predicted.
- Gold 3 (Severe): 30% <= FEV<sub>1</sub> (%) <50% predicted.
- Gold 4 (Very serious): FEV<sub>1</sub> (%) <30% predicted.

In case the number of GOLD 4 subjects was less than 10, these will be grouped with the GOLD 3 subjects, forming a single category (GOLD 3-4).

## 7.2.9 BODEx Index

The BODEx index includes the body mass index (BMI), the degree of dyspnea measured with the mMRC scale, the pulmonary function measured with the FEV<sub>1</sub> (%) post-bronchodilation and the

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

number of severe exacerbations (only visits to hospital emergencies and admissions are included). It is a continuous variable with a range from 0 to 9 points.

Table A: Calculation of the BODEx Index for prognostic approach to COPD.

| | Variables | Score | | | |
|----|-----------------------|-------|-------|-------|-----|
| | | 0 | 1 | 2 | 3 |
| В | BMI (kg/m2) | >21 | ≤21 | | |
| О | FEV <sub>1</sub> (%) | ≥65 | 50-64 | 36-49 | ≤35 |
| D | Dyspnea (mMRC)* | 0-1 | 2 | 3 | 4 |
| Ex | Severe Exacerbations) | 0 | 1-2 | ≥3 | |

Propuesto por (Soler-Cataluna et al. 2009)

Taking into account the score obtained in the BODEX index, they can be grouped into the following categories:

• Class I Mild: BODEx 0-2 points

• Class II Moderate: BODEx 3-4 points

• Class III Serious: BODEx 5-6 points

• Class IV Very serious: BODEx 7-9 points

## **7.2.10 COTE Index**

The COTE comorbidity index was constructed from the 12 comorbidities that were associated with a statistically significant risk of death (Divo et al. 2012). Thus, comorbidities such as hypertension and hypercholesterolemia, which are very frequent in patients with COPD, would not be associated with higher mortality, while others would be, such as cancer (particularly lung, esophagus, pancreas and breast), anxiety, liver cirrhosis, atrial fibrillation, diabetes, pulmonary fibrosis, heart failure, gastroduodenal ulcer and coronary heart disease.

The sum of the points aims to capture the individual or combination of diseases that affect each patient. The total score ranges between 0 and 25 points. An increase of 1 point in the COTE index is associated with an increased risk of death from episodes related to COPD and not related to COPD.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Table B: Comorbidities associated with mortality and the COTE index

| Disease | Points |
|--------------------------------------------|----------------------------|
| Lung, esophagus, pancreas or breast cancer | 6 |
| Pulmonary fibrosis | 2 |
| Auricular Fibrillation / flutter | 2 |
| Congestive heart failure | 1 |
| Coronary artery disease | 1 |
| Gastroduodenal ulcer | 1 |
| Liver cirrhosis | 2 |
| Diabetic neuropathy | 2 |
| Anxiety | 6 |
| All other cancers | 2 |
| Total score | $\sum$ (sum of all points) |

The COTE index will also be described according to the mortality risk at this cut-off point:

- Low risk mortality: COTE index <4 points
- High risk mortality: COTE index  $\geq$  4 points.

#### 7.2.11 Risk stratification

Patients will be classified according to their risk based on GesEPOC 2017 Spanish guideline:

- Low risk:
  - $\circ$  FEV<sub>1</sub>(%) post-bronchodilation >= 50% and,
  - o mMRC 0-2, and
  - o 0 or 1 exacerbation in the last year, and
  - o without hospitalization in the last year.
- High risk:
  - o FEV<sub>1</sub>(%) post-bronchodilation<50% or,
  - $\circ$  mMRC > 2 or mMRC = 2 with treatment or,
  - o 2 or more exacerbation in the last year or,
  - o 1 or more exacerbation with hospitalization in the last year.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 

#### 7.2.12 Gold 2019 Classification

According to GOLD 2019 classification, four different types of patients will be considered:

- Patient A:
  - o 0 or 1 exacerbations (not leading to hospital admission) and,
  - $\circ$  mMRC 0-1 and CAT < 10
- Patient B:
  - o 0 or 1 exacerbations (not leading to hospital admission), and
  - $\circ$  mMRC >= 2 or CAT >= 10
- Patient C:
  - $\circ \geq 2$  exacerbations or  $\geq 1$  exacerbation leading to hospital admission, and
  - $\circ$  mMRC 0-1 and CAT < 10.
- Patient D:
  - ≥2 exacerbations or any >= 1 exacerbation leading to hospital admission, and
  - $\circ$  mMRC >= 2 or CAT >= 10.

## 7.2.13 CAT questionnaire score

The CAT questionnaire score will be obtained from the sum of the 8 items that each range from 0 (no symptoms) to 5 points (highest symptoms) (Available at http://www.catestonline.org/).

Table C: CAT questionnaire and responses

| Item | Symptom | 0 option | Range | 5 option |
|---|---|---|---|---|
| 1 | Cough | I never cough | [0 5] | I cough all the time |
| 2 | Mucus | I have no phlegm (mucus) in my chest at all | [0 5] | My chest is completely full of phlegm (mucus) |
| 3 | Chest pressure | My chest does not feel tight at all | [0 5] | My chest feels very tight |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

| Item | Symptom | 0 option | Range | 5 option |
|---|---|---|---|---|
| 4 | Dyspnea | When I walk up a hill or one flight of stairs I am not breathless | [0 5] | When I walk up a hill or one flight of stairs I am very breathless |
| 5 | Limitation in domestic activities | I am not limited doing any activities at home | [0 5] | I am very limited doing activities at home |
| 6 | Social limitation | I am confident leaving my home despite my lung condition | [0 5] | I am not at all confident leaving my home because of my lung condition |
| 7 | Sleep | I sleep soundly | [0 5] | I don't sleep soundly because of my lung condition |
| 8 | Energy | I have lots of energy | [0 5] | I have no energy at all |
| | TOTAL | | [0-40] | |

Missing or missing answers are not allowed to obtain a valid score. Therefore, the score range of this questionnaire ranges from 0 to 40 points. The score will be grouped into two categories:

- CAT <10: Low impact of COPD (Most days are good, the illness prevents the patient from doing one or two things he or she would like, coughing several days a week).
- CAT  $\geq$ 10: Medium / high impact of COPD in the patient.

On the other hand, the CAT score will be categorized according to the impact of symptoms such as cough, mucus, chest pressure, dyspnea, limitation in domestic activities, social limitation and sleep and energy:

Low impact:  $0 \le CAT \le 10$ .

Moderate impact:  $11 \le CAT \le 20$ .

High impact: 21 <= CAT <= 30.

Very high impact:  $31 \le CAT \le 40$ .

#### Adherence to ICS treatment recommendations according GesEPOC 2017 guideline. 7.2.14

GESEPOC 2017 guideline indicates different treatment options according to risk and COPD Phenotype, obtained from Figure 4 in "Guía española de la enfermedad pulmonar obstructiva crónica (GesEPOC) 2017. Tratamiento farmacológico en fase estable" in

http://www.archbronconeumol.org/es-pdf-S0300289617300844.

\bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS Document: OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx

Author: Version Number:

1.0


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

The use of ICS is indicated only in these cases:

- Patients at high risk and,
  - OPD asthma syndrome (ACOS). Only mixed phenotype allows the use of ICS as the first option. For exacerbator with chronic bronchitis and exacerbator with emphysema, the use of ICS is indicated after a first treatment of LAMA / LABA, when there is worsening of symptoms.

Table D: Treatment COPD scheme according to risk and phenotype



Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015



Figure 4 in "Guía española de la enfermedad pulmonar obstructiva crónica (GesEPOC) 2017. Tratamiento farmacológico en fase estable" (http://www.archbronconeumol.org/es-pdf-S0300289617300844)

Taking into account the algorithm of treatment recommendations included in GesEPOC (phenotype) guidelines, we will define patients as:

- Adherent to ICS (Adequate use of ICS):
  - Patients treated with ICS that according to GesEPOC guidelines should have been treated with ICS, or
  - Patients **not** treated with ICS that according to GesEPOC guidelines should **not** have been treated with ICS.
- Non-Adherent to ICS (Inadequate use of ICS):
  - Patients treated with ICS but according to GesEPOC guidelines should **not** have been treated with ICS, or
  - Patients **not** treated with ICS but according to GesEPOC guidelines should have been treated with ICS.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 

#### 7.3 Software Version

All analyses will be conducted using SAS version 9.4. Other statistical packages that can be used are SPSS version 19.0 or higher.

## 8. STATISTICAL CONSIDERATIONS

## 8.1 Statistical Bias Reduction

Methods for handling bias will be discussed in the appropriate section for endpoints relating to missing values.

#### 8.2 Statistical Tests and Confidence Intervals

Unless otherwise specified in the description of the analyses, a two-sided 95% confidence interval will be considered as a default (alpha = 5%). P-values are provided as descriptive representations of the data, since no confirmatory testing is planned.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

8.3 Adjustments for Covariates and Factors to be Included in Analyses

For some of the endpoints, multivariate analyses will be performed using the following covariates and factors. For details of their inclusion in the models, see the specific analysis section. Fixed variables are:

• Age

Gender

Some optional variables are:

• Smoking history

• Number of exacerbations in the previous year.

• FEV<sub>1</sub> (%) or COPD severity

• FVC (%)

COPD Risk

• COPD Phenotype

• Gold 2019 Classification A, B, C, D

• Comorbidities as asthma and/or atopy

CAT category

8.4 Missing data

Missing data will not be imputed, except in those variables described in their scoring system.

According to general analysis, if patients have missing values for an outcome, those patients will be excluded for that outcome's analysis.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 

# 9. OUTPUT PRESENTATIONS

Tables and Figures on page 39 describe the presentations for this study and therefore the format and content of the summary TLFs to be provided by

RWES Biostatistics.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Statistical Analysis Plan Template 

10. DISPOSITION AND WITHDRAWALS

All subjects who provide informed consent will be accounted for in this study. Subject disposition,

withdrawals, and protocol violations (as defined in section 6.2), including inclusion and exclusion

criteria will be presented for all enrolled patients.

11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the FAS. General statistical

testing will be carried out for demographic or other baseline characteristics.

The following demographic and other baseline characteristics will be reported for this study:

• Age in study visit

Sex

• Ethnicity

• Weight (kg), Height (cm), Body mass index (BMI) (kg/m<sup>2</sup>) and categories

• Tobacco use (no-smoker, ex-smoker, smoker, packs/year)

• Time since diagnosis (years) - calculated relative to date of visit

11.1 Derivations

Derived variables are specified in section 7.2. Common Calculations on page 15 in this SAP.

12. SURGICAL AND MEDICAL HISTORY

Neither surgical nor medical history are collected in the eCRF.

13. COMORBIDITIES

Comorbidities are collected according to COTE index, plus asthma and athopy. Comorbidities will be presented for the FAS.

\bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Document:

## 14. MEDICATIONS

Medications will be presented for the FAS and coded using the WHO Drug Dictionary (WHO-DD) and Anatomical Therapeutic Chemical (ATC) class coding (including ATC Level 3).

Medications (antibiotics and corticosteroids) used for exacerbations, will be considered only if start date is in the two years previous to the study visit. Medications started previously will not be considered for analysis due to the exacerbations are not included in the study period.

## 15. STUDY MEDICATION EXPOSURE

Patients in this study will have been prescribed a treatment for their COPD. They could have been prescribed ICS or not. Prescription of the treatments will have been done under the sole responsibility of the healthcare professional and before the study initiation visit.

#### 16. PRIMARY OUTCOMES

#### 16.1 Primary Endpoint

The primary endpoint for a patient, currently on ICS, is absence or presence of moderate/severe exacerbation in the year prior to the study visit.

#### 16.1.1 Data Variables and Derivation

The data will be obtained from medical charts and it will be collected in "treatments" section (all treatment combinations including ICS will be considered as "yes" and also ICS discontinuation the same date of the study visit will be considered as "yes"). Treatments have to be started previously to the study visit and it have to be ongoing or stopped the same day of the study visit.

#### 16.1.2 Missing Data Methods for Primary Endpoint

Missing data will not be imputed. If patients have missing values for this outcome, those patients will be excluded for the analysis and number of missing values will be presented.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

16.1.3 Primary Analysis of Primary Endpoints

The primary analysis will consist of the proportion of patients, currently on ICS, who did not have or

had moderate/severe exacerbation in the year prior to the study visit. The primary analysis will be

performed for the FAS.

16.1.3.1 Current treatment with ICS

Main variable will be presented according to the presence or not of moderate/severe exacerbations in

the previous 365 days.

The use of ICS will be analyzed using number of patients in each category and percentages (absolute

and relative frequencies) and 95% confidence intervals will be provided based on Wald's (Normal

Approximation) method for each group. Percentages will be compared using Chi-Square test or

Fisher's Exact test.

Logistic regression will be used to assess the independent contribution of clinical and demographic

factors to the estimation of the proportion of patients with COPD who use ICS inadequately. First,

univariate and second, multiple logistic regression (MLR) methods will be used to investigate the

impact of the following explanatory covariates (patient and disease characteristics) on ICS use.

Potential covariates are:

Age

gender

Smoking history

• Number of exacerbations in the previous year.

• History of asthma (yes/no)

• History of atopy (yes/no)

COTE index

COPD GesEPOC 2017 phenotype

\\bcnfs02\general\\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\\8. SRO ESTUDIOS\\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Document:

• GOLD 2019 spirometric classifications (1, 2,3, 4)

• GOLD 2019 patient groups (A, B, C, D)

mMRC score

CAT - COPD Assessment Test

Backward selection procedures will be applied to generate the final MLR models which consider only covariates in the selection procedure with a p-value <0.1 in the corresponding univariate logistic regression analysis, using inadequate ICS use (yes/no) as response variable. A p-value <0.05 will be used for the covariates to stay in the model in a backward elimination step. Continuous variables can be replaced by categorical variables. Parameters estimated, exp(B) and C95% Wald Confidence Limits for OR will be presented.

Additionally, logistic regression model will be performed for each age subgroup, using the same procedure described in the previous paragraph. Age subgroups will be adjusted according to the distribution of patients.

## 16.1.3.2 Inadequate use of ICS

As a part of main analysis, inadequate use of ICS will be presented as in the previous section 16.1.3.1. Current treatment with ICS. This analysis will be presented only for patients without exacerbations in the previous year. This cohort will be used because only patients without exacerbations can receive ICS without requiring it, which is, making an inappropriate use of the treatment

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Statistical Analysis Plan Template 

#### 16.2 Secondary analysis

The secondary analyses will be performed for the FAS. According to previous statements, if patients have missing values for an outcome, those patients will be excluded for that outcome's analysis.

#### 16.2.1 ICS use in the two years prior to the study visit

The secondary analyses is the proportion of patients with COPD treated with ICS at the time of study visit with or without moderate-to-severe exacerbations, in the previous 2 years before the study visit (see also section 16.1.1. Data Variables and Derivation on page 29).

This analysis will be presented according to the presence or not of moderate/severe exacerbations in the previous 2x365 days.

Use of ICS will be analyzed using number of patients in each category and percentages (absolute and relative frequencies) and 95% confidence intervals will be provided based on Wald's (Normal Approximation) method for each group. Percentages will be compared using Chi-Square test or Fisher's Exact test.

#### 16.2.2 Moderate-to-severe exacerbations in COPD

This analysis consists of the number (count) of moderate-to-severe exacerbations in the previous 1 and 2 years previous to the study visit in COPD patients according to ICS use at time of study visit.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Patients with missing data related to exacerbations will be excluded from the analysis and number of missing values will be presented.

The objective is to describe the number (total count) of moderate-to-severe exacerbations in one and two years previous to the study visit according to ICS treatment at the time of study visit.

Results will be analyzed with measures of central tendency (mean and median), variability/dispersion (standard deviation and interquartile ranges) and ranges. The number of moderate-to-severe exacerbations will be analyzed using Mann-Whitney U test or Kruskal-Wallis non-parametric tests.

After that, at exploratory level, negative binomial regressions will be used for modelling discrete-count variables, not continuous and limited to non-negative values as the number of moderate-to-severe exacerbations (counts), both for first and second previous years. Covariates included in the model will be those used also in primary analysis, excluding the number of exacerbations in the previous year.

Backward selection procedures will be applied to generate the final model which consider only covariates in the selection procedure with a p-value <0.1 in the corresponding univariate analysis, using number of exacerbations as response variable. A p-value <0.05 will be used for the covariates to stay in the model in a backward elimination step. Continuous variables can be replaced by categorical variables.

## 16.2.3 General patient profile for COPD patients

To evaluate general patient profile for COPD patients, several variables will be described. In general, descriptive statistics will be used for describing the patient profile. All results will be analyzed with measures of central tendency (mean and median), variability/dispersion (standard deviation and interquartile ranges and ranges) for continuous variables and distributions of absolute and relative frequencies for categorical variables. This analysis will be also performed for the FAS.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

All results will be described according to the ICS treatment in the study visit: categorical variables will be analyzed using Chi-Square or Fisher's Exact test and quantitative variables by means t-test for independent groups or for quantitative variables that do not meet parametric applicability criteria, adequate statistical analysis will be used, as Mann-Whitney U test or Kruskal Wallis test. Variables included are:

Table 2. Variables included in the eCRF

| Group | Variable |
|---|---|
| Sociodemographic | Age (years), |
| | gender, |
| | ethnicity. |
| | BMI (Kg/m2) |
| | BMI grade |
| | Smoking history. |
| Clinical Variables | Spirometry - Bronchodilator test |
| | Spirometry - FEV1 absolute values pre and post-bronchodilator |
| | Spirometry - FEV1 % values pre and post-bronchodilator. |
| | Spirometry - FEV1 increase from pre to post-bronchodilator |
| | Blood Eosinophilia (number of eosinophils and %) |
| | Immunoglobulin E (Ig E) |
| Exacerbations | Episodes of exacerbations in the previous year |
| | Episodes of exacerbations in the two previous years |
| | Episodes of severe exacerbations in the previous year |
| | Episodes of severe exacerbations in the two previous years |
| | Treatments for exacerbations |
| COPD characteristics | Time since COPD diagnosis (years) |
| | COPD GesEPOC 2017 phenotypes |
| | GOLD 2019 spirometric classifications (Gold 1, Gold 2, Gold 3, Gold 4). |
| | GOLD 2019 patient groups (A, B, C, D). |
| | BODEx index (numerical and categories) |
| | Risk classification according GesEPOC. |
| | Breathlessness based on mMRC score. |
| | CAT - COPD Assessment Test (numerical and categories) |
| Comorbidities | COTE index (numerical and categories) |
| | History of asthma (yes/no) |
| | Time since asthma diagnosis (years) |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

| Group | Variable |
|---|---|
| | History of atopy (yes/no). |
| | Current COPD treatment: With ICS: ICS, LABA+ICS, LABA+LAMA+ICS. Without ICS: SABA, SAMA, LABA, LAMA, LABA+LAMA, Others |
| | History of antibiotics for COPD |
| | History of corticosteriods for COPD |
| | Concomitant medication. |
| | Adherence to GesEPOC 2017 treatment recommendations guidelines |

#### 16.2.4 Rescue medication use

The description of Rescue medication used in patients treated with ICS and without ICS will include the active substance (ATC codes), dose, start date and end date. The main treatment is salbutamol (SABA) and it will be described the number and percentage of patients who used each treatment as rescue medication in the last year and in the last two years. This percentage will be calculated using as denominator FAS set.

Results will be stratified by ICS treatment in the study visit. Percentages will be compared using Chi-Square or Fisher's Exact test.

#### 16.2.5 Adherence to GesEPOC 2017 treatment recommendations guidelines

Adherence to treatment recommendations according GesEPOC 2017 guidelines will be described using number and percentage of adherent patients (considered treated according to guidelines).

Tables will be described according to the number of exacerbations in the last year prior to study visit:

- patients with 0-1 exacerbations (not leading to hospital admission) vs.
- patients with ≥ 2 exacerbations or ≥ 1 exacerbation leading to hospital admission in the last 1 year;

Comparisons between groups will be performed using Chi-Square or Fisher's Exact test.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

#### 16.2.6 ICS-related adverse events

Percentage of patients treated with ICS who reported ICS-related events will be reported. All adverse event list will be presented (see Safety Outcomes).

## 17. PATIENT REPORTED OUTCOMES (PRO)

Quality of Life (QoL) was assessed using the COPD Assessment Test (CAT), a questionnaire for people with COPD designed to measure the impact of COPD on a person's life, and how these changes over time (http://www.catestonline.org/).

The analysis of CAT is included in analysis of patient profile in section 16.2.3. General patient profile for COPD patients (page 33).

#### 18. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the Safety Analysis Set (see sections 6.4 and 6.5).

#### 18.1 Adverse Drug Reactions

First of all, the percentage of patients experiencing ICS-related adverse drug reactions (ADRs) will be presented in patients using ICS. Only ADRs with onset date included in the last two years previous to study visit will be included.

Number and percentage of patients reporting each type of ADRs will be reported: Pneumonia, Fracture, Skin thinning/easy bruising, Cataract, Diabetes and Oropharyngeal candidiasis. ADRs will be described according to type, seriousness, reason for seriousness and outcome.

In the same way, the percentage of patients experiencing Adverse Drug Reactions related with BI products SPIOLTO®, STRIVERDI®, SPIRIVA® or ATROVENT® will be presented. Number and percentage of patients reporting each type of ADRs will be reported. ADRs will be described according to type, duration (days), seriousness, reason for seriousness and outcome.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015
Adverse Drug Reaction term (open string variable) will be coded using Medical Dictionary for

Regulatory Activities (MedDRA) central coding dictionary, Version 20.0.

**18.2** Serious Adverse Drug Reactions

Serious Adverse Drug Reactions (SADRs) are those ADRs recorded as "Serious" on the Adverse

Events page of the (e)CRF. A summary of serious SADRs by SOC and PT will be prepared.

The percentage of patients experiencing serious ICS-related adverse drug reaction (SADRs) will be

presented in patients using ICS. Only SADRs with onset date included in the last two years previous

to study visit will be included.

Number and percentage of patients reporting each type of SADRs will be reported: Pneumonia,

Fracture, Skin thinning/easy bruising, Cataract, Diabetes and Oropharyngeal candidiasis. Global

SADRs will be described according to type of seriousness and outcome.

The percentage of patients experiencing serious related drug reactions (SADRs) with SPIOLTO®,

STRIVERDI®, SPIRIVA® or ATROVENT® will be presented. Number and percentage of patients

reporting each type of SADRs will be reported.

18.3 Deaths

If any subjects die during ICS-treatment or SPIOLTO®, STRIVERDI®, SPIRIVA® or

ATROVENT® treatment, recorded on the "results in death" or outcome of event" as "fatal" on AEs

and ADRs page of the (e)CRF, the information will be presented in a summary table and a data

listing.

19. REFERENCES

Celli, B. (2017). Is the Blood Eosinophil Count a Useful Biomarker in COPD? The devil is in the

Details! Arch Bronconeumol 53(8): 415-416.

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Cosio, B. G., J. B. Soriano, J. L. Lopez-Campos, M. Calle-Rubio, J. J. Soler-Cataluna, J. P. de-Torres, J. M. Marin, C. Martinez-Gonzalez, P. de Lucas, I. Mir, G. Peces-Barba, N. Feu-Collado, I. Solanes, I. Alfageme, and C. Casanova. 2016. 'Defining the Asthma-COPD Overlap Syndrome in a COPD Cohort', Chest, 149: 45-52.

Divo, M., C. Cote, J. P. de Torres, C. Casanova, J. M. Marin, V. Pinto-Plata, J. Zulueta, C. Cabrera, J. Zagaceta, G. Hunninghake and B. Celli (2012). "Comorbidities and risk of mortality in patients with chronic obstructive pulmonary disease." Am J Respir Crit Care Med 186(2): 155-161.

Miravitles, M. (2015). Frequency and characteristics of different clinical phenotypes of chronic obstructive pulmonary disease. Int J Tuberc Lung Dis, Aug; 19(8) 992-8.

#### 19.1 Dated & Times

Depending on data available, dates and times will take the form <dd/mm/yyyy hh:mm:ss.>

## 19.2 Spelling Format

English UK.

### 19.3 Listings

All listings will be ordered by the following: group (ICS/non-ICS, etc..), center-subject ID, and date (where applicable).

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

## 20. TABLES AND FIGURES

## 20.1 Evaluability

### Table 3. Evaluability criteria – Patients in the FAS

| | | Total |
|------------------------------------|--------------------------|-------|
| Total included patients (ENR) | | |
| Evaluable patients | Evaluable patients (FAS) | |
| | Non-Evaluable patients | |
| Reasons for non-evaluable patients | Inclusion criteria 1 | |
| | Inclusion criteria 2 | |
| ICS Analysis Set (PICAS) | | |
| Safety Analysis Set-ICS | | |
| Safety Analysis Set- BI drug | | |

### Table 4. Other protocol violations occurred in evaluable patients

| | | Total |
|---|---|---|
| Evaluable patients | Evaluable patients (FAS) | |
| Important protocol violations | ADR (serious or non-serious) or fatal event not notified to BI | |
| | Any other major or critical Non-<br>Compliance detected during monitoring<br>visit | |

Table 5. Main stratification variables

| | | Total |
|---|---|---|
| Total evaluable (FAS) | | |
| Current treatment on ICS | Total No (Non - ICS treatment) Yes (ICS treatment) 95% CI for current ICS treatment | |
| Moderate/severe exacerbations in the previous year | Total No (Without Moderate/severe Exacerbations) Yes (With Moderate/severe Exacerbations) 95% CI for presence of moderate/severe exacerbations in the previous year | |
| Inadequate use of ICS | Total Adherent patients: Adequate use of ICS | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its

| | Total |
|---|---|
| Non-adherent patients: Inadequate use of ICS (use of ICS in patients without moderate/severe exacerbatic previous year) 95% CI for non-adherent patients (inadequate use of ICS) | ons in the |

## 20.2 General patient profile for COPD patients according to ICS current use

Main analysis will be stratified by current ICS treatment (patients currently treated with ICS vs. patients currently non-treated with ICS). The same tables for general patient profile could be presented according to GOLD (I-IV), GOLD (A-D) and GesEPOC Phenotypes.

### 20.2.1 Socio-demographic characteristics

Table 6. Socio-demographic variables and habits according to current treatment on ICS.

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Age | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Age group | 40-49 years<br>50-59 years<br>60-69 years<br>70-79 years<br>80+ years | | | |
| Gender | Male, n (%)<br>Female, n (%) | | | |
| Ethnicity | Caucasian<br>Asian<br>African<br>Unknown<br>Other | | | |
| Weight (Kg) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| | N missings | | | |
| Height (cm) | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missings | | | |
| BMI (Kg/m2) | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missings | | | |
| BMI cat | Underweight: BMI< 18.5 kg/m2 Normal weight: 18.5 kg/m2<= BMI<= 25 kg/m2 Overweight: 25 kg/m2< BMI<= 30 kg/m2 Obese: 30 kg/m2 <bmi<= 35="" bmi="" kg="" m2="" obese:="" severely=""> 35 kg/m2</bmi<=> | | | |
| Smoking habit | Non-smoker<br>Smoker<br>Ex-smoker | | | |
| Smokers-<br>Number of years smoking | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| Smokers-<br>Number of pack-years | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| Ex-Smokers-<br>Number of years smoking | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| Ex-Smokers-<br>Number of pack-years | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

Document:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its

### 20.2.2 Clinical variables

Table 7. Spirometry values in COPD patients according to current treatment on ICS.

| | | | Non - ICS | ICS | Total |
|---|---|---|---|---|---|
| Pre-bronchodilator | FVC (L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FVC (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1 (L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1 (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1/FVC (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Post-bronchodilator | FVC (L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FVC (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1 (L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1 (%) | Valid N | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | | Non - ICS | ICS | Total |
|---|---|---|---|---|---|
| | | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1/FVC (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1/FVC (%) - cat | FEV1/FVC (%) < 0.7<br>FEV1/FVC (%) ≥ 0.7 | | | |
| Change | FEV1 Change (L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1 percentage of change (1) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | FEV1 percentage of change (2) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

Table 8. Comorbidities according to current treatment on ICS.

| | | Non - ICS | ICS | Total |
|-----------------------------|--------------------|-----------|-----|-------|
| History of asthma | No | | | |
| | Yes | | | |
| Time since asthma diagnosis | Valid N | | | |
| (years) | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| History of atopy | No | | | |
| | Yes | | | |
| COTE Index -comorbidities | Lung cancer | | | |
| | Esophagus cancer | | | |
| | Pancreas cancer | | | |
| | Breast cancer | | | |
| | Pulmonary fibrosis | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| | Auricular Fibrillation / flutter Congestive heart failure Coronary artery disease Gastroduodenal ulcer Liver cirrhosis Diabetic neuropathy Anxiety All other cancers | | | |
| COTE Index | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| COTE Index (cat) | Low risk: COTE index <4 points<br>High risk: COTE index ≥ 4 points. | | | |

Table 9. COPD characteristics according to current treatment on ICS.

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Time since COPD diagnosis (years) | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| Time since COPD diagnosis (cat) | 0-2 years<br>>2-5 years<br>>5 years | | | |
| COPD GesEPOC<br>2017 phenotypes | non-exacerbator,<br>mixed COPD - asthma syndrome (ACOS)<br>exacerbator with emphysema<br>exacerbator with chronic bronchitis | | | |
| GOLD 2019<br>spirometric classification | Gold 1 – Mild<br>Gold 2 – Moderate<br>Gold 3 – Severe<br>Gold 4 – Very severe | | | |
| GOLD 2019 patient groups (A, B, C, D). | Patient A Patient B Patient C Patient D | | | |
| BODEx Index | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| BODEx Index (cat) | Class I Mild: BODEx 0-2 points Class II Moderate: BODEx 3-4 points Class III Serious: BODEx 5-6 points Class IV Very serious: BODEx 7-9 points | | | |
| CAT score | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| CAT score (cat) | CAT <10: Low impact of COPD. CAT ≥10: Medium / high impact of COPD Low impact: 0 <= CAT <= 10. Moderate impact: 11 <= CAT <= 20. High impact: 21 <= CAT <= 30. Very high impact: 31 <= CAT <= 40. | | | |
| mMRC score | Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 | | | |

Table 10. Analytic results according to current treatment on ICS.

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Blood Eosinophilia (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Number of eosinophils (%) | <2%<br>>= 2% | | | |
| Blood Eosinophilia (cel/μl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Number of eosinophils (cel/μl) | <100 cel/μl<br>100-299 cel//μl<br>>= 300 cel/μl | | | |
| Immunoglobulin E (UI/ml) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| | N missing | | | |
| Inmunoglobulin E (UI/ml) | ≤100 UI/ml<br>>100 UI/ml | | | |

### 20.2.3 Exacerbations

Table 11. Previous exacerbations according to current treatment on ICS.

| Period | Variable | | Non - ICS | ICS | Total |
|---|---|---|---|---|---|
| Last 2 years | Total Exacerbations | No<br>Yes | | | |
| | Number of total Exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | Moderate/Severe Exacerbations | No<br>Yes | | | |
| | Number of Moderate/Severe<br>Exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | Severe Exacerbations | No<br>Yes | | | |
| | Number of Severe Exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Previous year | Total Exacerbations | No<br>Yes | | | |
| | Number of total Exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| | Moderate/Severe Exacerbations | No<br>Yes | | | |
| | Number of Moderate/Severe<br>Exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3) | | | |

Document:

\\bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| Period | Variable | | Non - ICS | ICS | Total |
|---|---|---|---|---|---|
| | | Min-Max<br>N missing | | | |
| | Severe Exacerbations | No<br>Yes | | | |
| | Number of Severe Exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

Table 12. Treatments for Moderate/Severe Exacerbations according to current treatment on ICS.

| | | Non - ICS | ICS | Total patients with severe/moderate exacerbations |
|---|---|---|---|---|
| Treatments for exacerbations | No<br>Yes | | | |
| Type of treatment (multirresponse) | Antibiotics for COPD β-Lactam antibiotics Amoxicillin/Clavulanic Acid Other Macrolides Azithromycin Other Fluoroquinolones Ciprofloxacin Levofloxacin Moxifloxacin Other Unknown antibiotic | | | |
| | Oral corticosteriods for COPD Systemic corticosteroids Prednisone Prednisolone Metilprednisolone Dexamethasone Deflazacort Other systemic corticosteroid Other Corticosteroid Unknown corticosteroid | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

### 20.2.4 Current COPD treatment

Table 13. Current COPD treatment according to current treatment on ICS

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| ICS treatment | No ICS<br>ICS alone<br>LABA + ICS<br>LABA + LAMA + ICS | 100% | 0% | |
| Type of ICS | ICS alone Budesonide Fluticasone propionate | -<br>-<br>- | | |
| | LABA + ICS Beclometasone / Formoterol Formoterol / Budesonide Salmeterol / Fluticasone propionate Fluticasone furoate/vilanterol LABA + LAMA + ICS | -<br>-<br>-<br>- | | |
| | Fluticasone / Umeclidinium / Vilanterol<br>Beclometasone / Formoterol / Glycopyrronium | - | | |
| Other treatments | No<br>Yes | | | |
| Type of treatment (multirresponse) | Inhaled therapy SABA Salbutamol Terbutaline SAMA Ipratropium LABA Formoterol Salmeterol Indacaterol Olodaterol LAMA Tiotropium Aclidinium Glycopyrronium Umeclidinium LABA+LAMA Indacaterol / Glycopyrronium Aclidinium / Formoterol Umeclidinium / Vilanterol Tiotropium / Olodaterol Other therapies | | | |
| | PDE4 inhibitors Roflumilast | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Non - ICS | ICS | Total |
|-----------------------------|-----------|-----|-------|
| Methylxanthines | | | |
| Theophylline | | | |
| Mucolytics | | | |
| Ambroxol | | | |
| Bromhexine | | | |
| Erdosteine | | | |
| Carbocisteine | | | |
| N-Acetylcysteine | | | |
| Other mucolytic | | | |
| Vaccines | | | |
| Influenza | | | |
| Conjugated pneumococcal | | | |
| Non-conjugated pneumococcal | | | |
| Antitussives | | | |
| Alpha-1-Antitrypsin | | | |
| Immunoregulators | | | |
| Other treatment | | | |

Percentages will be calculated over total of patients in each group (100%).

Table 14. Presentation of current COPD treatment pattern according to current treatment on ICS

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| ICS alone | | - | | |
| Budesonide | □ TH: 100 mcg/inh □ TH: 200 mcg/inh □ TH: 400 mcg/inh | - | | |
| Fluticasone propionate | □ PCI: 50 mcg/inh □ PCI: 125 mcg/inh □ PCI: 250 mcg/inh □ AH: 100 mcg/inh □ AH: 250 mcg/inh □ AH: 500 mcg/inh | - | | |
| LABA + ICS | | - | | |
| Beclometasone / Formoterol | □ NH: 100/6 mcg/inh □ PCI Modulite: 100/6 mcg/inh | - | | |
| Formoterol / Budesonide | □ TH: 4,5/160 mcg/inh □ TH: 9/320 mcg/inh □ SM: 4,5/160 mcg/inh □ SM: 9/320 mcg/inh □ EH: 4,5/160 mcg/inh □ EH: 9/320 mcg/inh | - | | |
| Salmeterol / Fluticasone propionate | □ AH: 50/500 mcg/inh □ FP: 50/500 mcg/inh | - | | |
| Fluticasone furoate/vilanterol | □ EL: 100/25 mcg/inh | - | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| LABA + LAMA + ICS | | - | | |
| Fluticasone / Umeclidinium / Vilanterol | □ EL: 92/65/22 mcg/inh | - | | |
| Beclometasone / Formoterol / Glycopyrronium | □ PCI: 87/5/9mcg/inh | - | | |
| Inhaled therapy | | | | |
| SABA | | | | |
| Salbutamol | □ PCI: 100mcg/inh | | | |
| Terbutaline | □ TH: 500 mcg/inh | | | |
| SAMA | | | | |
| Ipratropium | □ PCI: 20mcg/inh | | | |
| LABA | | | | |
| Formoterol | □ PCI: 12 mcg/inh | | | |
| | □ TH: 9 mcg/inh □ AL: 12mcg/inh | | | |
| Salmeterol | □ PCI: 25 mcg/inh | | | |
| Sameteror | □ AH: 50 mcg/inh | | | |
| Indacaterol | □ BH: 150mcg/inh | | | |
| | □ BH: 300 mcg/inh | | | |
| Olodaterol | □ RM: 2,5 mcg/inh | | | |
| LAMA | | | | |
| Tiotropium | □ HA: 18 mcg/inh □ RM: 2,5 mcg/inh | | | |
| Aclidinium | □ GE: 400 mcg/inh | | | |
| Glycopyrronium | □ BH: 44 mcg/inh | | | |
| Umeclidinium | □ EL: 62,5 mcg/inh | | | |
| LABA+LAMA | | | | |
| Indacaterol / Glycopyrronium | □ BH: 110/50 mcg/inh | | | |
| Aclidinium / Formoterol | □ GE: 340/12 mcg/inh | | | |
| Umeclidinium / vilanterol | □ EL: 62,5/25 mcg/inh | | | |
| Tiotropium / Olodaterol | □ RM: 2,5/2,5mcg/inh | | | |
| - | | | | |
| Other therapies | | | | |
| PDE4 inhibitors | | | | |
| Roflumilast | □ 250 mcg/tablet □ 500 mcg/tablet | | | |
| Metilxantines | | | | |
| Theophylline | □ 100 retard mg/tablet □ 200 retard mg/tablet □ 300 retard mg/tablet □ Oral Solution 27mg/5ml | | | |
| Mucolytics | | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Ambroxol | □ Oral Solution 15mg/5ml □ Oral Solution 300mg/100ml □ Tablets 30 mg | | | |
| Bromhexine | □ Oral Solution 160mg/100ml □ Oral Solution 80mg/100ml □ Tablets 8mg | | | |
| Erdosteine | □ Oral Solution 3,5g/100ml □ Tablets 300 mg | | | |
| Carbocisteine | □ Oral Solution 50mg/100ml □ Oral Solution 100mg/ml □ Sachets: 750mg | | | |
| N-Acetylcysteine | □ Sachets 200mg □ Sachets 600mg | | | |
| Other mucolytic | | | | |

Percentages (each presentation) will be calculated over the patients receiving each treatment.

Table 15. Doses of current COPD treatment pattern according to current treatment on ICS

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| ICS alone | | - | | |
| Budesonide | 200-1600 mcg/24h | - | | |
| | mcg/ h | | | |
| | mcg/ h Not available | | | |
| Fluticasone propionate | 500 mcg/12h | - | | |
| | mcg/ h | | | |
| | mcg/ h | | | |
| | Not available | | | |
| LABA + ICS | | - | | |
| Beclometasone / Formoterol | 200/12 mcg/12h | - | | |
| | / mcg/ h | | | |
| | / mcg/ h | | | |
| | Not available | | | |
| Formoterol / Budesonide | 9/320 mcg/12h | - | | |
| | / mcg/ h | | | |
| | / mcg/ h<br>Not available | | | |
| Salmeterol / Fluticasone propionate | 50/500 mcg/12h | - | | |
| | / mcg/ h | | | |
| | / mcg/ h | | | |
| | Not available | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

<sup>\*</sup> AH: Accuhaler; AL: Aerolizer; BH: Breezhaler; IC: Inhaled capsules; EH: Easyhaler; EL: Ellipta; FP: Forspiro; GE: Genuair; HA: Handihaler; IPC: Inhaler in pressurized cartridge; inh: inhalation; NT: Nexthaler; RM: Respimat; SM: Spiromax; TH: Turbuhaler.

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Fluticasone furoate/vilanterol | 100/25 mcg/24h<br>XX1/YY1 mcg/ZZ1 h<br>XX2/YY2 mcg/ZZ2 h<br>Not available | - | | |
| LABA + LAMA + ICS | | - | | |
| Fluticasone / Umeclidinium / Vilanterol | 92/65/22 mcg/24h// mcg/ h// mcg/ h Not available | - | | |
| Beclometasone / Formoterol / Glycopyrronium | 2 inhal 87/5/9 mcg/ 12h<br>_// mcg/ h<br>_//_ mcg/ h<br>Not available | - | | |
| Inhaled therapy | | | | |
| SABA | | | | |
| Salbutamol | 200 mcg/4-6h mcg/ h mcg/ h Not available | | | |
| Terbutaline | 500 mcg/6h mcg/ h mcg/ h Not available | | | |
| SAMA | | | | |
| Ipratropium | 20-40 mcg/6-8h mcg/ h mcg/ h Not available | | | |
| LABA | | | | |
| Formoterol | 12 mcg/12h mcg/ h mcg/ h Not available | | | |
| Salmeterol | 50 mcg/12h mcg/ h mcg/ h Not available | | | |
| Indacaterol | 150 mcg/24h mcg/ h mcg/ h Not available | | | |
| Olodaterol | 5 mcg/24h<br>mcg/ h<br>mcg/ h<br>Not available | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| LAMA | | | | |
| Tiotropium | 18 mcg/24h 05 mcg/24h mcg/ h mcg/ h Not available | | | |
| Aclidinium | 400 mcg/12h mcg/ h mcg/ h Not available | | | |
| Glycopyrronium | 44 mcg/24h mcg/ h mcg/ h Not available | | | |
| Umeclidinium | 62,5 mcg/24h mcg/ h mcg/ h Not available | | | |
| LABA+LAMA | | | | |
| Indacaterol / Glycopyrronium | 110/50 mcg/24h/ mcg/ h/ mcg/ h Not available | | | |
| Aclidinium / Formoterol | 340/12 mcg/12h/ mcg/ h/ mcg/ h Not available | | | |
| Umeclidinium / vilanterol | 62,5/25 mcg/24h/ mcg/ h/_ mcg/ h Not available | | | |
| Tiotropium / Olodaterol | 5/5 mcg/24h/ mcg/ h/ mcg/ h Not available | | | |
| Other therapies | | | | |
| PDE4 inhibitors | | | | |
| Roflumilast | 250-500 mcg/24h mcg/ h mcg/ h Not available | | | |
| Metilxantines | | | | |
| Theophylline | 400 mg/24h mg/ h mg/ h | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| | Not available | | | |
| Mucolytics | | | | |
| Ambroxol | 30 mg/8h mg/ h mg/ h Not available | | | |
| Bromhexine | 8 mg/8h mg/ h mg/ h Not available | | | |
| Erdosteine | 300 mg/12h mg/ h mg/ h Not available | | | |
| Carbocisteine | 750 mg/8h mg/ h mg/ h Not available | | | |
| N-Acetylcysteine | 200 mg/8h mg/ h nd h Not available | | | |
| Other mucolytic | mg/ h mg/ h Not available | | | |
| Vaccines | | | | |
| Influenza | | | | |
| Conjugated pneumococcal | | | | |
| Non-conjugated pneumococcal | | | | |
| Antitussives | mg/ h mg/ h Not available | | | |
| Alpha-1-Antitrypsin | mg/ h mg/ h Not available | | | |
| Immunoregulators | mg/ h mg/ h Not available | | | |
| Other treatment | | | - | |

Percentages (each dose) will be calculated over the patients receiving each treatment.

Table 16. Time in treatment (months) of current COPD treatment pattern according to current treatment on ICS

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| ICS alone | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Budesonide | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Fluticasone propionate | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| LABA + ICS | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Beclometasone / Formoterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Formoterol / Budesonide | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Salmeterol / Fluticasone propionate | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Fluticasone furoate/vilanterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| LABA + LAMA + ICS | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Fluticasone / Umeclidinium / Vilanterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Beclometasone / Formoterol / Glycopyrronium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | - | | |
| Inhaled therapy | | | | |
| SABA | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Salbutamol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Terbutaline | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| SAMA Document: | Mean (SD)<br>Median (Q1-Q3) | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| | Min-Max | | | |
| Ipratropium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| LABA | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Formoterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Salmeterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Indacaterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Olodaterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| LAMA | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Tiotropium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Aclidinium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Glycopyrronium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Umeclidinium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| LABA+LAMA | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Indacaterol / Glycopyrronium | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Aclidinium / Formoterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Umeclidinium / vilanterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Tiotropium / Olodaterol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Other therapies | | | | |
| PDE4 inhibitors | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Roflumilast | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Metilxantines | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Theophylline | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Mucolytics | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Ambroxol | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Bromhexine | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Erdosteine | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Carbocisteine | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| N-Acetylcysteine | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Other mucolytic | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Vaccines | | | | |
| Influenza | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Conjugated pneumococcal | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Non-conjugated pneumococcal | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Antitussives | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Alpha-1-Antitrypsin | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Immunoregulators | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Other treatment | | | | |

### 20.2.5 Previous COPD treatment

Table 17. Previous COPD treatment according to current treatment on ICS

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Previous 2 years | No ICS<br>ICS alone<br>LABA + ICS<br>LABA + LAMA + ICS | | | |
| | ICS alone Budesonide Fluticasone propionate | | | |
| | LABA + ICS Beclometasone / Formoterol Formoterol / Budesonide Salmeterol / Fluticasone propionate Fluticasone furoate/vilanterol | | | |
| | LABA + LAMA + ICS Fluticasone / Umeclidinium / Vilanterol Beclometasone / Formoterol / Glycopyrronium | | | |
| Last year | No ICS<br>ICS alone<br>LABA + ICS<br>LABA + LAMA + ICS | | | |
| | ICS alone Budesonide Fluticasone propionate | | | |
| | LABA + ICS Beclometasone / Formoterol Formoterol / Budesonide | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Non - ICS | ICS | Total |
|---|---|---|---|
| Salmeterol / Fluticasone propionate<br>Fluticasone furoate/vilanterol | | | |
| LABA + LAMA + ICS Fluticasone / Umeclidinium / Vilanterol Beclometasone / Formoterol / Glycopyrronium | | | |

Percentages will be calculated over total of patients in each group (100%).

Table 18. Presentation of previous COPD treatment according to current treatment on ICS

| | | Presentation | Group1 | Group2 | Total |
|---|---|---|---|---|---|
| Previous 2 years | ICS alone | | | | |
| | Budesonide | □ TH: 100 mcg/inh □ TH: 200 mcg/inh □ TH: 400 mcg/inh | | | |
| | Fluticasone propionate | □ PCI: 50 mcg/inh □ PCI: 125 mcg/inh □ PCI: 250 mcg/inh □ AH: 100 mcg/inh □ AH: 250 mcg/inh □ AH: 500 mcg/inh | | | |
| | LABA + ICS | | | | |
| | Beclometasone / Formoterol | □ NH: 100/6 mcg/inh □ PCI Modulite: 100/6 mcg/inh | | | |
| | Formoterol / Budesonide | □ TH: 4,5/160 mcg/inh □ TH: 9/320 mcg/inh □ SM: 4,5/160 mcg/inh □ SM: 9/320 mcg/inh □ EH: 4,5/160 mcg/inh □ EH: 9/320 mcg/inh | | | |
| | Salmeterol / Fluticasone propionate | □ AH: 50/500 mcg/inh □ FP: 50/500 mcg/inh | | | |
| | Fluticasone furoate/vilanterol | □ EL: 100/25 mcg/inh | | | |
| | LABA + LAMA + ICS | | | | |
| | Fluticasone / Umeclidinium / Vilanterol | □ EL: 92/65/22 mcg/inh | | | |
| | Beclometasone / Formoterol / Glycopyrronium | □ PCI: 87/5/9mcg/inh | | | |
| Last year | ICS alone | | | | |
| | Budesonide | □ TH: 100 mcg/inh □ TH: 200 mcg/inh □ TH: 400 mcg/inh | | | |
| | Fluticasone propionate | □ PCI: 50 mcg/inh | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Presentation | Group1 | Group2 | Total |
|---|---|---|---|---|
| | □ PCI: 125 mcg/inh □ PCI: 250 mcg/inh □ AH: 100 mcg/inh □ AH: 250 mcg/inh □ AH: 500 mcg/inh | | | |
| LABA + ICS | | | | |
| Beclometasone / Formoterol | □ NH: 100/6 mcg/inh □ PCI Modulite: 100/6 mcg/inh | | | |
| Formoterol / Budesonide | □ TH: 4,5/160 mcg/inh □ TH: 9/320 mcg/inh □ SM: 4,5/160 mcg/inh □ SM: 9/320 mcg/inh □ EH: 4,5/160 mcg/inh □ EH: 9/320 mcg/inh | | | |
| Salmeterol / Fluticasone propionate | □ AH: 50/500 mcg/inh □ FP: 50/500 mcg/inh | | | |
| Fluticasone furoate/vilanterol | □ EL: 100/25 mcg/inh | | | |
| LABA + LAMA + ICS | | | | |
| Fluticasone / Umeclidinium / Vilanterol | □ EL: 92/65/22 mcg/inh | | | |
| Beclometasone / Formoterol / Glycopyrronium | □ PCI: 87/5/9mcg/inh | | | |

Percentages (each presentation) will be calculated over the patients receiving each treatment.

Table 19. Doses of previous COPD treatment according to current treatment on ICS

| | | Doses | Group1 | Group2 | Total |
|---|---|---|---|---|---|
| Previous 2 | ICS alone | | | | |
| years | Budesonide | 200-1600 mcg/24h mcg/ h mcg/ h Not available | | | |
| | Fluticasone propionate | 500 mcg/12h mcg/ h mcg/ h Not available | | | |
| | LABA + ICS | | | | |
| | Beclometasone / Formoterol | 200/12 mcg/12h<br>/ mcg/ h<br>/ mcg/ h<br>Not available | | | |
| | Formoterol / Budesonide | 9/320 mcg/12h<br>/ mcg/ h<br>/ mcg/ h | | | |

Document:

\\bcnfs02\general\\Hdmgener\\MEDICAL AFFAIRS 28.02.2017 actualizada\\8. SRO ESTUDIOS\\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Doses | Group1 | Group2 | Total |
|---|---|---|---|---|---|
| | | Not available | | | |
| | Salmeterol / Fluticasone propionate | 50/500 mcg/12h<br>/ mcg/ h<br>/ mcg/ h<br>Not available | | | |
| | Fluticasone furoate/vilanterol | 100/25 mcg/24h<br>XX1/YY1 mcg/ZZ1 h<br>XX2/YY2 mcg/ZZ2 h<br>Not available | | | |
| | LABA + LAMA + ICS | | | | |
| | Fluticasone / Umeclidinium / Vilanterol | 92/65/22 mcg/24h// mcg/ h/_/ mcg/ h Not available | | | |
| | Beclometasone / Formoterol / Glycopyrronium | 2 inhal 87/5/9 mcg/ 12h<br>/_/ mcg/ h<br>/_/ mcg/ h<br>Not available | | | |
| Last year | ICS alone | | | | |
| Last year | Budesonide | 200-1600 mcg/24hmcg/hmcg/h Not available | | | |
| | Fluticasone propionate | 500 mcg/12h<br>mcg/ h<br>mcg/ h<br>Not available | | | |
| | LABA + ICS | | | | |
| | Beclometasone / Formoterol | 200/12 mcg/12h<br>/ mcg/ h<br>/_ mcg/ h<br>Not available | | | |
| | Formoterol / Budesonide | 9/320 mcg/12h/ mcg/ h/_ mcg/ h Not available | | | |
| | Salmeterol / Fluticasone propionate | 50/500 mcg/12h<br>_/ mcg/ h<br>_/_ mcg/ h<br>Not available | | | |
| | Fluticasone furoate/vilanterol | 100/25 mcg/24h<br>XX1/YY1 mcg/ZZ1 h<br>XX2/YY2 mcg/ZZ2 h<br>Not available | | | |
| | LABA + LAMA + ICS | | | | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | Doses | Group1 | Group2 | Total |
|---|---|---|---|---|
| Fluticasone / Umeclidinium / Vilanterol | 92/65/22 mcg/24h/_/ mcg/ h/_/ mcg/ h Not available | | | |
| Beclometasone / Formoterol / Glycopyrronium | 2 inhal 87/5/9 mcg/ 12h<br>/_/ mcg/ h<br>/_/ mcg/ h<br>Not available | | | |

Percentages (each dose) will be calculated over the patients receiving each treatment.

### 20.2.6 Rescue medication

Table 20. Use and type of rescue medication in the previous 2 years according to current treatment on ICS

| | | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Use of rescue medication | No<br>Yes<br>Not available in Clinical records | | | |
| Rescue medication | SABA (salbutamol) Other treatments Treatment 1 Treatment 2 | | | |
| Time (days) with salbutamol<br>Within 2 years | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Time (days) with Treatment 1 * Within 2 years | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |

Percentages will be calculated over total of patients in each group (100%). (\*): If there is a high number of other rescue medication, time in treatment will be analyzed for each medication.

Table 21. Use and type of rescue medication in the previous year according to current treatment on ICS

| | | Group1 | Group2 | Total |
|---|---|---|---|---|
| Use of rescue medication | No<br>Yes<br>Not available in Clinical records | | | |
| Rescue medication | SABA (salbutamol) | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Group1 | Group2 | Total |
|---|---|---|---|---|
| | Other treatments Treatment 1 Treatment 2 | | | |
| Time (days) with salbutamol<br>Within previous year | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |
| Time (days) with Treatment 1 * Within previous year | Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | |

Percentages will be calculated over total of patients in each group (100%). (\*): If there is a high number of other rescue medication, time in treatment will be analyzed for each medication.

## 20.2.7 Concomitant treatments (ATC code classification)

Table 22. Concomitant treatments according to current treatment on ICS

| | Doses | Non - ICS | ICS | Total |
|---|---|---|---|---|
| Other treatments | No<br>Yes | | | |
| Type of treatment | A Alimentary tract and metabolism A10 Drugs used in diabetes A10B Blood glucose lowering drugs, excl. insulins A10BA Biguanides A10BA01 Phenformin A10BA02 Metformin A10BA03 Buformin N Nervous System. N02 Analgesics. N02B Other analgesics and antipyretics. N02BE Anilides. N02BE01 Paracetamol (acetaminophen). N02BE01 Paracetamol N02BE03 Phenacetin N02BE04 Bucetin N02BE05 Propacetamol | | | |

Percentages will be calculated over total of patients in each group (100%).

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Table 23. Comorbidities (receiving treatment) according to current treatment on ICS

| Doses | Non - ICS | ICS | Total |
|---------------------------------------|-----------|-----|-------|
| Total Comorbidity 001 Comorbidity 002 | | | |

Percentages will be calculated over total of patients in each group (100%).

## 20.3 Endpoints

#### 20.3.1 ICS treatment

Table 24. Current treatment on ICS according to the absence or presence of moderate/severe exacerbations in the year prior to the study visit.

| ICS treatment | Moderate/severe Exacerbations in the previous year | | Total |
|---|---|---|---|
| | No | No Yes | |
| Total patients | N (100%) | N (100%) | N (100%) |
| Currently non treated with ICS | XXX (XX.X%)<br>[95%CI: XX.X%-XX.X] | XXX (XX.X%)<br>[95%CI: XX.X%-XX.X] | XXX (XX.X%)<br>[95%CI: XX.X%-XX.X] |
| Currently treated with ICS | XXX (XX.X%)<br>[95%CI: XX.X%-XX.X] | XXX (XX.X%)<br>[95%CI: XX.X%-XX.X] | XXX (XX.X%)<br>[95%CI: XX.X%-XX.X] |

<sup>\*</sup>Note: Percentages will be column percentages. Each percentage will correspond to percentage of patients currently treated with ICS, according to the presence of moderate/severe exacerbations in the previous year.

Table 25. Inadequate use of ICS (use of ICS without moderate/severe exacerbations in the previous year) according to clinical and demographic factors (univariate logistic regression analysis)

| Variable | Category | • | Odds-Ratio<br>(OR) | p-value |
|---|---|---|---|---|
| Age | Cont (1 year) | n/N (%) | | |
| | 40-49 years<br>50-59 years<br>60-69 years<br>70-79 years<br>80+ years | n/N (%)<br>n/N (%)<br>n/N (%)<br>n/N (%)<br>n/N (%) | (ref) | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| Variable | Category | Inadequate use of ICS | Odds-Ratio<br>(OR) | p-value |
|---|---|---|---|---|
| Gender | Male<br>Female | | (ref) | |
| BMI cat | Underweight: BMI< 18.5 kg/m2 Normal weight: 18.5 kg/m2<= BMI<= 25 kg/m2 Overweight: 25 kg/m2< BMI<= 30 kg/m2 Obese: 30 kg/m2 <bmi<= 35="" bmi="" kg="" m2="" obese:="" severely=""> 35 kg/m2</bmi<=> | | (ref) | |
| Smoking habit | Non-smoker<br>Smoker<br>Ex-smoker | | (ref) | |
| History of asthma | No<br>Yes | | (ref) | |
| History of atopy | No<br>Yes | | (ref) | |
| BODEx Index (cat) | Class I Mild: BODEx 0-2 points<br>Class II Moderate: BODEx 3-4 points<br>Class III Serious: BODEx 5-6 points<br>Class IV Very serious: BODEx 7-9 points | | (ref) | |
| COTE Index (cat) | Low risk: COTE index <4 points<br>High risk: COTE index ≥ 4 points. | | (ref) | |
| Time since COPD diagnosis (cat) | 0-2 years >2-5 years >5 years | | (ref) | |
| COPD GesEPOC<br>2017 phenotypes | non-exacerbator,<br>mixed COPD - asthma syndrome (ACOS),<br>exacerbator with emphysema<br>exacerbator with chronic bronchitis | | (ref) | |
| GOLD 2019<br>spirometric classification | Gold 1 – Mild<br>Gold 2 – Moderate<br>Gold 3 – Severe<br>Gold 4 – Very severe | | (ref) | |
| GOLD 2019 patient groups (A, B, C, D) | Patient A Patient B Patient C Patient D | | (ref) | |
| CAT score (cat) | CAT <10: Low impact of COPD.<br>CAT ≥10: Medium / high impact of COPD | | (ref) | |
| mMRC score | Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 | | (ref) | |
| Number of eosinophils (%) | <2%<br>>= 2% | | (ref) | |


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| <= 100 UI/ml<br>>100 UI/ml | | (maf) | |
|---|---|---|---|
| | | (ref) | |
| None 1-2 exacerbations 3-4 exacerbations 5+ exacerbations | | (ref) | |
| None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations | | (ref) | |
| None 1-2 severe exacerbations 3-4 severe exacerbations 5+ severe exacerbations | | (ref) | |
| None 1-2 exacerbations 3-4 exacerbations 5+ exacerbations | | (ref) | |
| None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations | | (ref) | |
| None 1-2 severe exacerbations 3-4 severe exacerbations 5+ severe exacerbations | | (ref) | |
| No<br>Yes | | (ref) | |
| No<br>Yes | | (ref) | |
| ICS alone<br>LABA + ICS<br>LABA + LAMA + ICS | | | |
| | 3-4 exacerbations 5+ exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations None 1-2 severe exacerbations 3-4 severe exacerbations 5+ severe exacerbations None 1-2 exacerbations 3-4 exacerbations 5+ exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations 1-2 severe exacerbations None 1-2 severe exacerbations 1-3 severe exacerbations 1-4 severe exacerbations 1-5 severe exacerbations 1-5 severe exacerbations 1-2 severe exacerbations 1-2 severe exacerbations 1-3 severe exacerbations 1-4 severe exacerbations 1-5 severe exacerbations 1-5 severe exacerbations 1-6 severe exacerbations 1-7 severe exacerbations 1-8 severe exacerbations 1-9 severe exacerbations 1-1 severe exacerbations 1-2 severe exacerbations 1-3 severe exacerbations 1-4 severe exacerbations 1-5 severe exacerbations | 3-4 exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations None 1-2 severe exacerbations 3-4 severe exacerbations 5+ severe exacerbations None 1-2 exacerbations 3-4 exacerbations 5+ exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations None 1-2 severe exacerbations 1-2 severe exacerbations None 1-2 severe exacerbations 1-2 severe exacerbations None 1-2 severe exacerbations 1-2 severe exacerbations 1-3 severe exacerbations No Yes No Yes ICS alone LABA + ICS | 3-4 exacerbations 5+ exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations None 1-2 severe exacerbations 3-4 severe exacerbations None 1-2 exacerbations None 1-2 exacerbations 3-4 exacerbations 3-4 exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations S+ severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations None 1-2 severe exacerbations S+ severe exacerbations S- severe exacerbations S- severe exacerbations S- severe exacerbations No Yes No Yes ICS alone LABA + ICS |

Inadequate use of ICS: use of ICS without moderate/severe exacerbations in the previous year in patients.

# Table 26. Multivariate logistic regression model of inadequate use of ICS (use of ICS without moderate/severe exacerbations in the previous year)

| Parameter | Cat | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > ChiSq | Exp(Est) |
|---|---|---|---|---|---|---|---|
| Intercept | | | | | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its

| Parameter | Cat | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > ChiSq | Exp(Est) |
|---|---|---|---|---|---|---|---|
| Variable 1 | | | | | | | |
| Variable 2 | Cat 2<br>Cat 3<br>Cat 4 | | | | | | |
| Variable n | | | | | | | |

| Effect | OR<br>Point Estimate | 95% Wald<br>Confidence Limits |
|------------|----------------------|-------------------------------|
| Variable 1 | | |
| Variable 2 | | |
| Variable n | | |

# Table 27. Multivariate logistic regression model of inadequate use of ICS (use of ICS without moderate/severe exacerbations in the previous year) by age subgroups

| | Patients age<br>years | | Patients aged | l xx- xx years | | | Patients age<br>years | |
|---|---|---|---|---|---|---|---|---|
| Effect | OR (95% CI) | p-value | OR (95% CI) | OR (95% CI) | OR (95% CI) | p-value | OR (95% CI) | p-value |
| Variable 1 | | | | | | | | |
| Variable 2 | | | | | | | | |
| Variable n | | | | | | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018


### 20.3.2 Exacerbations

Statistical Analysis Plan Template

Table 31. Presence of moderate/severe exacerbations in COPD patients in the year previous to the study visit according to current treatment on ICS

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|---|
| Number of moderate/severe exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Presence of moderate/severe exacerbations | Total Without exacerbations With exacerbations | | | |
| | None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations | | | |

# Table 32. Negative binomial model for number of moderate-to-severe exacerbations in COPD patients in the year previous to the study visit

| Parameter | DF | Estimate | Std Error | Wal 95% CI | Chi-Square | Pr>ChiSq |
|------------|----|----------|-----------|------------|------------|----------|
| Variable 1 | | | | | | |
| Variable 2 | | | | | | |
| Variable n | | | | | | |
| Dispersion | | | | | | |

# Table 33. Presence of total exacerbations in COPD patients in the year previous to the study visit according to current treatment on ICS

| | | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|---|
| Number of total exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Presence of exacerbations | Total Without exacerbations With exacerbations None | | | |
| | 1-2 exacerbations | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its

| | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|
| 3-4 exacerbations<br>5+ exacerbations | | | |

# Table 34. Presence of severe exacerbations in COPD patients in the year previous to the study visit according to current treatment on ICS

| | | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|---|
| Number of severe exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Presence of severe exacerbations | Total Without exacerbations With exacerbations | | | |
| | None 1-2 exacerbations 3-4 exacerbations 5+ exacerbations | | | |

# Table 35. Presence of moderate/severe exacerbations in COPD patients in the two previous years to the study visit according to current treatment on ICS

| | | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|---|
| Number of moderate/severe exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Presence of moderate/severe exacerbations | Total Without exacerbations With exacerbations | | | |
| | None 1-2 moderate/severe exacerbations 3-4 moderate/severe exacerbations 5+ moderate/severe exacerbations | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| on treated with ICS | Currently treated with ICS | Total |
|---------------------|----------------------------|-------|

# Table 36. Presence of total exacerbations in COPD patients in the two previous years to the study visit according to current treatment on ICS

| | | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|---|
| Number of total exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Presence of exacerbations | Total Without exacerbations With exacerbations | | | |
| | None 1-2 exacerbations 3-4 exacerbations 5+ exacerbations | | | |

Table 37. Presence of severe exacerbations in COPD patients in the two previous years to the study visit according to current treatment on ICS

| | | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|---|
| Number of severe exacerbations | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missings | | | |
| Presence of severe exacerbations | Total Without exacerbations With exacerbations | | | |
| | None<br>1-2 exacerbations | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to Holdin subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its

| | Non treated with ICS | Currently treated with ICS | Total |
|---|---|---|---|
| 3-4 exacerbations<br>5+ exacerbations | | | |

## 20.3.3 Adherence to treatment recommendations according GesEPOC 2017 guidelines.

Table 38. Adherence to treatment recommendations according to GesEPOC 2017 Guidelines, according to number of exacerbations in the last year

| | | 0-1 * | >= 2 ** | Total |
|---|---|---|---|---|
| | | exacerbations | exacerbations | |
| Adherence | Adherent (Adequate ICS use) ICS-Treated who should be treated with ICS Non ICS-treated who should not be treated with ICS Non-Adherent (Non-adequate ICS use) ICS-Treated who should not be treated with ICS Non ICS-treated who should be treated with ICS | | | |

<sup>\* 0-1</sup> exacerbations (not leading to hospital admission). \*\*  $\geq$  2 exacerbations or  $\geq$  1 exacerbation leading to hospital admission in the last 1 year prior to index date.

### 20.4 Safety

## 20.4.1 Adverse Drug Reactions - related with ICS

Table 39. Patients with ADRs related with ICS treatment according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| ADRs related with ICS treatment | Total Patients<br>No<br>Yes | | | |
| Type of ADR (multi-response) | <ul><li>□ Pneumonia</li><li>□ Fracture</li><li>□ Skin thinning/easy bruising</li></ul> | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Current<br>Non - ICS | Current<br>ICS | Total<br>ICS patients |
|---|---|---|---|---|
| | □ Cataract □ Diabetes □ Oropharyngeal candidiasis | | | |
| ADR outcome (multi-response) | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with ICS at some time during the previous two years.

Table 40. Description of ADRs related with ICS treatment according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| Number of ADRs related with ICS treatment | Total ADRs ICS-related | | | |
| Type of ADR | <ul> <li>□ Pneumonia</li> <li>□ Fracture</li> <li>□ Skin thinning/easy bruising</li> <li>□ Cataract</li> <li>□ Diabetes</li> <li>□ Oropharyngeal candidiasis</li> </ul> | | | |
| ADR outcome | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with ICS at some time during the previous two years

Table 41. List of ADRs related with ICS treatment

| PATCOD | Adverse Event Term | MedDRA Code | Onset date | End<br>date | SAE? | Reason for seriousness | Outcome |
|---|---|---|---|---|---|---|---|

Patients in the Safety Analysis Set. Including patients treated with ICS at some time during the previous two years

\\bcnfs02\general\\Hdmgener\\MEDICAL AFFAIRS 28.02.2017 actualizada\\8. SRO ESTUDIOS\\RESPIRATORIO\1237-0070 NIS Document:

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its


## 20.4.2 Serious Adverse Drug Reactions (SADRs) - related with ICS

Table 42. Patients with SADRs related with ICS treatment according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| SADRs related with ICS treatment | Total patients<br>No<br>Yes | | | |
| Type of SADR<br>(multi-response) | <ul> <li>□ Pneumonia</li> <li>□ Fracture</li> <li>□ Skin thinning/easy bruising</li> <li>□ Cataract</li> <li>□ Diabetes</li> <li>□ Oropharyngeal candidiasis</li> </ul> | | | |
| Reason for seriousness<br>(multi-response) | Results in death Immediately life-threatening Persistent or significant disability/incapacity Requires/prolongs hospitalization Congenital anomaly/birth defect Other comparable medical criteria | | | |
| SADR outcome<br>(multi-response) | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with ICS at some time during the previous two years

Table 43. Description of SADRs related with ICS treatment according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| Number of SADRs related with ICS treatment | Total SADRs ICS-related | | | |
| Type of SADR | □ Pneumonia □ Fracture □ Skin thinning/easy bruising □ Cataract □ Diabetes □ Oropharyngeal candidiasis | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| Reason for seriousness | Results in death Immediately life-threatening Persistent or significant disability/incapacity Requires/prolongs hospitalization Congenital anomaly/birth defect Other comparable medical criteria | | | |
| SADR outcome | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with ICS at some time during the previous two years

# **20.4.3** Adverse Drug Reactions associated to BI product (SPIOLTO®, STRIVERDI®, SPIRIVA® or ATROVENT®)

Table 44. Patients with ADRs associated to BI product according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| ADRs associated to BI product | Total Patients<br>No<br>Yes | | | |
| Type of ADR (multi-response) | Term 1 Term 2 Term n | | | |
| ADR outcome<br>(multi-response) | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with BI product at some time during the previous two years.

Table 45. Description of ADRs associated to BI product according to current treatment on ICS

| | Current<br>Non - ICS | Current<br>ICS | Total<br>ICS patients |
|---|----------------------|----------------|-----------------------|
| · | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx

Y . D . [20] [A] [20]

Version Number:


Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Template No.: RWI\_TP\_BIOS0013 Revision 1

Author:

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its

1.0

| | | Current<br>Non - ICS | Current<br>ICS | Total<br>ICS patients |
|---|---|---|---|---|
| ADRs associated to BI product | Total ADRs | | | |
| Type of ADR | Term 1 Term 2 Term n | | | |
| ADR outcome | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with BI product at some time during the previous two years

Table 46. List of ADRs associated with BI product.

| PATCOD | Adverse Event Term | MedDRA Code | Onset date | Reason for seriousness | Relationship<br>With BI product |
|---|---|---|---|---|---|

Patients in the Safety Analysis Set. Including patients treated with BI product at some time during the previous two years

## 20.4.4 Serious Adverse Drug Reaction (SADRs)related with BI product

Table 47. Patients with SADRs related with BI product according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total<br>ICS patients |
|---|---|---|---|---|
| SADRs associated to BI product | Total patients<br>No | | | |

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

| | | Current<br>Non - ICS | Current<br>ICS | Total<br>ICS patients |
|---|---|---|---|---|
| | Yes | | | |
| Type of SADR (multi-response) | Term 1 Term 2 Term n | | | |
| Reason for seriousness<br>(multi-response) | Results in death Immediately life-threatening Persistent or significant disability/incapacity Requires/prolongs hospitalization Congenital anomaly/birth defect Other comparable medical criteria | | | |
| SADR outcome<br>(multi-response) | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with BI product at some time during the previous two years

Table 48. Description of SADR related with BI product according to current treatment on ICS

| | | Current<br>Non - ICS | Current<br>ICS | Total ICS patients |
|---|---|---|---|---|
| Number of SADRs associated to BI product | Total SADRs | | | |
| Type of SADR | Term 1 Term 2 Term n | | | |
| Reason for seriousness | Results in death Immediately life-threatening Persistent or significant disability/incapacity Requires/prolongs hospitalization Congenital anomaly/birth defect Other comparable medical criteria | | | |
| SADR outcome | Recovered Not yet recovered Recovered with secuelae Unknown Fatal | | | |

Patients in the Safety Analysis Set. Including patients treated with BI product at some time during the previous two years

Document: \bcnfs02\general\Hdmgener\MEDICAL AFFAIRS 28.02.2017 actualizada\8. SRO ESTUDIOS\RESPIRATORIO\1237-0070 NIS

OPTI\11 - Clinical Trial Report\SAP\SAP - V 1.0\SAP OPTI version1.0 29052019.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Holdings Inc. and its


### **20.4.5** Deaths

#### Table 49. List of deaths

| PATCOD | Adverse Event Term | MedDRA Code | Onset date | End date | Outcome | Relationship<br>With BI product |
|---|---|---|---|---|---|---|

Document:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018